CLINICAL TRIAL: NCT01542294
Title: Phase I/II Study of Oral S-1 Plus f Oxaliplatin as an Adjuvant Chemotherapy After Curative Resection of Stage II-IV(M0) Gastric Cancer
Brief Title: SOX as Adjuvant Chemotherapy for Resectable Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Lin Yang, associated professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-020
Record Dates: First submitted 2011-10-16; First posted 2012-03-02 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; S-1; oxaliplatin; adjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); titanium silicide; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): s1+oxaliplatin
  Interventions: Drug: s1; Drug: Oxaliplatin

INTERVENTIONS:
Drug: s1 — 60-90mg/m2/d P.O. day 1-14, repeated every 21 days
  Other Names: TS-1
Drug: Oxaliplatin — 130mg/m2 d1 repeated every 21 days
  Other Names: Eloxatin

SUMMARY:
The purpose of this study is to assess the safety and efficacy of S-1 plus oxaliplatin combination chemotherapy based on the adverse events and survival period by performing a phase I/II study of this combination in patients with D2 resection of gastric cancer.

DETAILED DESCRIPTION:
This stage I/II study is designed to evaluate the appropriate dose of S-1 plus fixed-dose of oxaliplatin (SOX regimen) for Patients with D2 resection of gastric cancer and survival of SOX regimen for stage II-III patients(AJCC 7th). To assess the efficacy, data on recurrence and survival will be collected from the time of enrollment until 3 years after surgery. To evaluate safety, data on adverse events will be collected from the time of enrollment until 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 20-70 years
* Histologically proven adenocarcinoma of the stomach
* Curative D2 lymphadenectomy resection for gastric cancer, who can start chemotherapy be within 6 weeks after surgery
* Stage II, III (AJCC 7th edition)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* No prior chemotherapy or radiotherapy
* Adequate bone marrow, renal, and liver function

Exclusion Criteria:

* Any evidence of metastatic disease (including presence of tumor cells in the ascites).
* Previous cytotoxic chemotherapy, radiotherapy or immunotherapy except corticosteroids, for the currently treated gastric cancer.
* Major surgery within 4 weeks prior to study treatment start, or lack of complete recovery from the effects of major surgery.
* Pregnant or lactating women.
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix.
* Lack of physical integrity of the upper gastrointestinal tract or those who have malabsorption syndrome likely to influence absorption of capecitabine, or inability to take oral medication.
* Organ allografts requiring immunosuppressive therapy.
* Serious uncontrolled intercurrent infections or other serious uncontrolled concomitant disease.
* Prior unanticipated severe reaction to fluoropyrimidine therapy (with or without documented dihydropyrimidine dehydrogenase (DPD) deficiency) or patients with known DPD deficiency. Hypersensitivity to platinum compounds or any of the components of the study medications.
* Received any investigational drug or agent/procedure, i.e. participation in another trial, within 4 weeks before enter the trial.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-06; Primary Completion 2014-09 (Actual); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
chemotherapy complete rate | 6 months
  percentage of patients who completed eight cycles of chemotherapy

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 years
  assessed from surgery until 1 months after withdrawing from study
recurrence-free survival(RFS) | 3 years
  from the date of surgery until the occurrence of an event (relapse or death whichever came first)
overall survival(OS) | 3 years
  from the date of surgery to any cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yang, MD, Principal Investigator — Department of Medical Oncology,Cancer Hospital and Institute,CAMS
Locations (1):
- Department of Medical Oncology,Cancer hospital and Institute,CAMS, Beijing, China

REFERENCES:
- [Derived] Wang G, Zhao J, Song Y, Zhang W, Sun Y, Zhou A, Huang J, Du F, Yang L. Phase II study of adjuvant chemotherapy with S1 plus oxaliplatin for Chinese patients with gastric cancer. BMC Cancer. 2018 May 9;18(1):547. doi: 10.1186/s12885-018-4480-9. PMID 29743043